CLINICAL TRIAL: NCT06883123
Title: Efficacy and Tolerability of Simbrinza and Rocklatan vs. Cosopt
Brief Title: Efficacy of Simbrinza and Rocklatan vs Cosopt and Latanoprost
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Prairie Eye Center (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: SY-25-01
Record Dates: First submitted 2025-03-12; First posted 2025-03-19 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — dorzolamide-timolol combination; Latanoprost; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Simbrinza and Rocklatan (Experimental): SIMBRINZA (brinzolamide and brimonidine tartrate) 1%/0.2% ROCKLATAN (netarsudil and latanoprost) 0.02%/0.005%
  Interventions: Drug: Simbrinza 0.2%-1% Ophthalmic Suspension; Drug: Rocklatan 0.02%-0.005% Ophthalmic Solution
- Cosopt and Latanoprost (Active Comparator): COSOPT (dorzolamide hydrochloride and timolol maleate) 2%/0.5% Latanoprost 0.005%
  Interventions: Drug: Cosopt PF 2%-0.5% Ophthalmic Solution; Drug: Latanoprost 0.005% Ophthalmic Solution

INTERVENTIONS:
Drug: Simbrinza 0.2%-1% Ophthalmic Suspension — brinzolamide and brimonidine tartrate
  Arms: Simbrinza and Rocklatan
Drug: Rocklatan 0.02%-0.005% Ophthalmic Solution — netarsudil and latanoprost
  Arms: Simbrinza and Rocklatan
Drug: Cosopt PF 2%-0.5% Ophthalmic Solution — dorzolamide hydrochloride and timolol maleate
  Arms: Cosopt and Latanoprost
Drug: Latanoprost 0.005% Ophthalmic Solution — Latanoprost
  Arms: Cosopt and Latanoprost

SUMMARY:
A randomized, multi-site, parallel-group, prospective study of patients who are adults with a diagnosis of mild to moderate open-angle glaucoma (OAG), currently on an on-label use of combination topical medication of Cosopt and Latanoprost for a minimum of 1 month.

ELIGIBILITY:
Inclusion criteria:

* Adults aged Eighteen (18) years and older with a diagnosis of mild to moderate open-angle glaucoma (OAG), currently on an on-label use of combination topical medication of Cosopt and Latanoprost for a minimum of 1 month. Evidence of optic nerve damage will be based on AAO Preferred Practice Patterns guidelines using either or both of the following:
* Optic disc or retinal nerve fiber layer (RNFL) structural abnormalities
* Diffuse or focal narrowing, or notching, of the optic disc rim, especially at the inferior or superior poles, which forms the basis for the ISNT rule
* Progressive narrowing of the neuroretinal rim with an associated increase in cupping of the optic disc
* Diffuse or localized abnormalities of the parapapillary RNFL, especially at the inferior or superior poles
* Disc rim, parapapillary RNFL, or lamina cribrosa hemorrhages
* Optic disc neural rim asymmetry of the two eyes consistent with loss of neural tissue
* Large extent of parapapillary atrophy
* Reliable and reproducible visual field abnormality considered a valid representation of the subject's functional status
* Visual field damage consistent with RNFL damage (e.g. nasal step, arcuate field defect, or paracentral depression in clusters of test sites)
* Visual field loss across the horizontal midline in one hemifield that exceeds loss in the opposite hemifield (in early/ moderate cases)
* Absence of other known explanations (e.g. optic disc drusen, optic nerve pit)
* Mean diurnal IOP ≥ 18 mmHg and < 28 mmHg at baseline in at least one eye with an inter-eye IOP difference < 5 mmHg.
* A central corneal thickness (CCT) within the range of 450-650 µm

Exclusion criteria:

* Patients with prior ocular procedures or intraocular surgery within 1 year prior to baseline (e.g. cataract surgery).
* Patients with prior history of glaucoma surgeries or laser treatment except patients with history of SLT >1 yr prior to baseline.
* Contraindications or known hypersensitivity to any or all the study medications including Rocklatan, Simbrinza, Cosopt and Latanoprost or related class of drugs.
* Patients with known history or presence of uncontrolled systemic diseases including diseases that, in investigator's opinion, may make it unsafe or undesirable for the subject to participate in the study and/ or limit adherence.
* Patients with known history or presence of significant ocular diseases including corneal diseases, dystrophies or abnormalities that would prevent accurate IOP readings with GAT.
* Patients with a history of uncontrolled IOP with the combination of either Rocklatan + Simbrinza or Cosopt + Latanoprost dual therapy.
* Significant ocular surface findings (e.g. hyperemia, irritation) found during slit lamp examination that might affect the study.
* Chronic use of any systemic medication for chronic diseases that may affect IOP.
* Subjects who are pregnant, lactating or planning a pregnancy.
* Any condition in the opinion in the investigator that would potentially confound the results of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Decrease in mean diurnal IOP | from baseline at week 8
  Mean diurnal IOP is determined as the average IOP measured at 8:30am, 12:00pm and 3:30pm

SECONDARY OUTCOMES:
Mean decrease in IOP at 8:30am | from baseline at week 8
Mean decrease in IOP at 12:00pm | from baseline at week 8
Mean decrease in IOP at 4:30pm | from baseline at week 8

OTHER OUTCOMES:
Mean % IOP diurnal reduction | from baseline at week 8
  Determined as the percentage decrease in average IOP measured at 8:30am, 12:00pm and 3:30pm

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Yeh, MD, Principal Investigator — Prairie Eye Center
Locations (1):
- Prairie Eye Center, Springfield, Illinois, United States

IPD SHARING:
Plan to Share IPD: No